CLINICAL TRIAL: NCT06411639
Title: A Multicenter, Open-label, Single-arm, Multiple-dose Study to Characterize the Pharmacokinetics, Safety and Tolerability of Subcutaneous Ianalumab in Chinese Adult Participants With Autoimmune Diseases
Brief Title: Pharmacokinetics Study of Ianalumab in Chinese Participants With Autoimmune Diseases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736A2104
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Sjogren Disease; Systemic Lupus Erythematosus
Keywords: Pharmacokinetic (PK); Systemic lupus erythematosus (SLE); Sjogren Disease (SjD); VAY736; ianalumab; B cell depletion
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — ianalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ianalumab 300 mg (Experimental): Participants will receive Ianalumab 300 mg subcutaneous (s.c.) monthly
  Interventions: Drug: ianalumab

INTERVENTIONS:
Drug: ianalumab — ianalumab will be provided in a pre-filled Syringe (PFS) of 150 mg/1 mL for s.c. administration. Two injections of 1mL each will be administered monthly.
  Other Names: VAY736

SUMMARY:
The purpose of this pharmacokinetic (PK) study is to describe the PK profile of ianalumab following s.c. administration in Chinese participants with systemic lupus erythematosus (SLE) and/or Sjögren's disease (SjD). Collection of intensive PK data from Chinese population had been designed in the ianalumab Phase 3 studies of SjD CVAY736A2302 (NCT05349214) and lupus nephritis (LN) CVAY736K12301 (NCT05126277) on an optional basis. This study is conducted to provide supplementary Chinese PK data in addition to the intensive PK data from the two Phase 3 studies .

DETAILED DESCRIPTION:
The study consists of the following periods:

* Screening Period: up to 4 weeks
* Treatment Period (Week 0 - Week 12) : 12 weeks
* Extended Treatment Period (after the completion of Week 12 - Week 52 (End of Treatment (EoT)) : 40 weeks

  ~ After completion of the 12-week treatment, participants will have the option to enter the Extended Treatment Period. If a participant does not enter the Extended Treatment Period, the EoT visit will be performed at the next planned visit following the completion of Week 12, followed by the Post-treatment Follow-up Period.
* Post-treatment Follow-up Period: at least 20 weeks and up to 2 years from the last dose of study treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients 18 years to 70 years of age (inclusive)
* Body weight at least 35 kg and not more than 120 kg and must have a body mass index (BMI) within the range of 18 - 35 kg/m2. BMI = Body weight (kg) / [Height (m)]2 at screening
* Diagnosed with SjD and/or SLE as determined by the investigator
* Have active disease (SjD and/or SLE) that may benefit from B-cell depletion therapy, as determined by the investigator.
* Participants currently receiving protocol-allowed SoC should be on stable doses of SoC medications for 4 weeks prior to first dosing of study treatment

Key Exclusion Criteria:

* Use of prohibited therapies
* Active viral, bacterial or other infections requiring systemic treatment at the time of screening or baseline or history of recurrent clinically significant infection
* Receipt of live/attenuated vaccine within a 4-week period before first dosing
* Uncontrolled co-existing serious disease
* Pregnant or nursing (lactating) women
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, refusing or unable to use highly effective methods of contraception while on study treatment and for 6 months after stopping of study drug

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-12-17 (Estimated); Study Completion 2028-06-24 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) calculated to the end of a dosing interval (tau) at steady-state (AUCtau) of ianalumab after the 3rd dose | Week 8 to 12 (Day 57): Pre-dose, Post-dose (24 hours (hr) +/- 12hr, 72 hr +/- 24 hr, 168 hr +/- 72 hr, 336 hr +/- 72hr, 504 hr +/- 72hr)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ianalumab. AUCtau of ianalumab will be summarized with descriptive statistics.
Observed maximum blood concentration (Cmax)of ianalumab after the 3rd dose | Week 8 to 12 (Day 57): Pre-dose, Post-dose (24 hours (hr) +/- 12hr, 72 hr +/- 24 hr, 168 hr +/- 72 hr, 336 hr +/- 72hr, 504 hr +/- 72hr)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ianalumab. Cmax of ianalumab will be summarized with descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) of ianalumab after the 3rd dose | Week 8 to 12 (Day 57): Pre-dose, Post-dose (24 hours (hr) +/- 12hr, 72 hr +/- 24 hr, 168 hr +/- 72 hr, 336 hr +/- 72hr, 504 hr +/- 72hr)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ianalumab. Tmax of ianalumab will be summarized with descriptive statistics.

SECONDARY OUTCOMES:
Ctrough of ianalumab at the end of dosing interval | Week 8 to 12 (Day 57): Pre-dose, Post-dose (24 hours (hr) +/- 12hr, 72 hr +/- 24 hr, 168 hr +/- 72 hr, 336 hr +/- 72hr, 504 hr +/- 72hr)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of ianalumab. Ctrough of ianalumab will be summarized with descriptive statistics.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | From date of enrollment till 30 days after end of Treatment, assessed up to approximately 44 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Anti-ianalumab antibodies (ADA) | Day 1 (Baseline), Week 8 to 11 Day 57 (Pre-dose), Week 12 Day 85, Week 24 Day 169, Week 36 Day 253, Week 52 Day 365, Week 68 Day 477 and Week 156 Day 1093
  Immunogenicity (IG) blood samples will be collected for anti-drug antibodies characterization. ADA of ianalumab will be summarized with descriptive statistics.
Presence of anti-drug antibodies (ADA) | Day 1 (Baseline), Week 8 to 11 Day 57 (Pre-dose), Week 12 Day 85, Week 24 Day 169, Week 36 Day 253, Week 52 Day 365, Week 68 Day 477 and Week 156 Day 1093
  Immunogenicity (IG) blood samples will be collected to assess the presence ADA of ianalumab.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No